CLINICAL TRIAL: NCT05221762
Title: Accelerated Cardiovascular Magnetic Resonance in Coronary Artery Disease
Brief Title: Accelerated Stress CMR in Coronary Artery Disease
Status: Active, not recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: University of Glasgow (Other); Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 0726; 258996 (Other: Health Research Authority)
Record Dates: First submitted 2021-11-15; First posted 2022-02-03 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Cardiovascular magnetic resonance (CMR) — Cardiovascular magnetic resonance (CMR) at 3 Tesla

SUMMARY:
This study will evaluate the diagnostic performance of an accelerated stress CMR protocol, comparing it with that of standard CMR assessment.

DETAILED DESCRIPTION:
This is a prospective, single-centre diagnostic accuracy study comparing the diagnostic performance of (1) accelerated and (2) standard adenosine stress CMR scans in 167 patients with suspected coronary artery disease referred for invasive coronary angiography (which will serve as the reference standard - invasive FFR).

The accelerated scan comprises accelerated cine and gadolinium imaging, with a standard stress scan (0.075mmol/kg gadolinium contrast).

Subjects will undergo both scans pre-angiography (in randomised order), enabling a head-to-head comparison of diagnostic performance (diagnostic accuracy, sensitivity and specificity) for identifying functionally significant coronary disease (as defined by fractional flow reserve <0.80).

Objectives The primary objective is to determine, in patients with suspected angina, whether the accelerated CMR protocol achieves favourable diagnostic accuracy, using invasive FFR as the reference standard, and also compared with standard CMR assessment.

Secondary objectives include comparing diagnostic performance of the accelerated CMR protocol with that of CT-FFR, a comparison of scan duration (overall and for each component - for standard and accelerated CMR), and patient tolerability and experience for each protocol (accelerated CMR, standard CMR and CTCA), as determined by a self-administered questionnaire rating patient comfort, symptoms experienced and perceived scan duration.

Data analysis

* Imaging data will be interpreted using the 16-segment American Heart Association (AHA) segmentation model
* For visual assessment of perfusion, images will be analysed by two experienced cardiologists, acting independently (differences resolved by consensus).
* For qualitative analysis, perfusion data will be analysed concurrently with late gadolinium images, with inducible ischaemia determined by the presence of a perfusion defect exceeding the area of scar.
* For quantitative analysis, myocardial blood flow (MBF) will be quantified using inline Gadgetron data (flow maps providing segmental flows).
* For qualitative analysis, ischaemia is defined as reversible hypoperfusion in two adjacent segments [32-segment model] exceeding the region of scar [if present], and for quantitative analysis, using a MBF threshold of 1.9ml/min/g.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Referred for invasive coronary angiography for investigation of chest pain
* Willing and able to give informed consent
* Willing and able (in the Investigators opinion) to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.
* Able to understand written English

Exclusion Criteria:

* Recent acute coronary syndrome (< 6 months)
* Severe claustrophobia
* Absolute contraindications to CMR - those with MR conditional or safe devices will be included
* Second-/third-degree atrioventricular block
* Severe chronic obstructive pulmonary disease
* Moderate-severe asthma
* Estimated glomerular filtration rate <30 ml/min/1.73m2
* Women who are pregnant, breast-feeding or of child-bearing potential (premenopausal women)
* Contraindication to iodinated contrast
* Participants who have participated in a research study involving an investigational product in the past 12 weeks
* Patients unable to understand written English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with suspected angina referred to Glenfield Hospital, Leicester, UK, for invasive coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of accelerated CMR (qualitative assessment) | 6 weeks
  Per vessel diagnostic accuracy of the accelerated CMR protocol (with qualitative perfusion assessment) and standard CMR protocol versus invasive coronary angiography with fractional flow reserve.
Diagnostic performance of accelerated CMR (quantitative assessment) | 6 weeks
  Per vessel diagnostic accuracy of the accelerated CMR protocol (with quantitative perfusion assessment) and standard CMR protocol versus invasive coronary angiography with fractional flow reserve.

SECONDARY OUTCOMES:
Sensitivity of accelerated CMR (vessel level) | 6 weeks
  Per vessel sensitivity of the accelerated protocol versus invasive coronary angiography with fractional flow reserve. This comparison will comprise two separate assessments of sensitivity against the reference standard - (1) algorithm with qualitative perfusion assessment (2) algorithm with quantitative perfusion assessment
Specificity of accelerated CMR (vessel level) | 6 weeks
  Per vessel specificity of the accelerated protocol versus invasive coronary angiography with fractional flow reserve. This comparison will comprise two separate assessments of specificity against the reference standard - (1) algorithm with qualitative perfusion assessment (2) algorithm with quantitative perfusion assessment
Sensitivity of accelerated CMR (patient level) | 6 weeks
  Per patient sensitivity of the accelerated protocol versus invasive coronary angiography with fractional flow reserve. This comparison will comprise two separate assessments of sensitivity against the reference standard - (1) algorithm with qualitative perfusion assessment (2) algorithm with quantitative perfusion assessment
Specificity of accelerated CMR (patient level) | 6 weeks
  Per patient specificity of the accelerated protocol versus invasive coronary angiography with fractional flow reserve. This comparison will comprise two separate assessments of specificity against the reference standard - (1) algorithm with qualitative perfusion assessment (2) algorithm with quantitative perfusion assessment
Diagnostic performance of accelerated CMR versus CTCA/FFRCT (1) | 6 weeks
  Per patient diagnostic accuracy of the accelerated CMR protocol (with qualitative perfusion assessment) for functionally significant coronary artery disease [CAD] (per patient level), compared with the diagnostic accuracy of CTCA/FFRCT.
Diagnostic performance of accelerated CMR versus CTCA/FFRCT (2) | 6 weeks
  Per patient diagnostic accuracy of the accelerated CMR protocol (with quantitative perfusion assessment) for functionally significant CAD (per patient level), compared with the diagnostic accuracy of CTCA/FFRCT.
Diagnostic performance of accelerated CMR versus computed tomography coronary angiography with computed tomography-derived fractional flow reserve (CTCA/FFRCT) (2) | 6 weeks
  Per patient diagnostic accuracy of the accelerated CMR protocol (with quantitative perfusion assessment) for functionally significant CAD (per patient level), compared with the diagnostic accuracy of CTCA/FFRCT.
Utility of rest perfusion assessment (1) | 6 weeks
  Diagnostic accuracy (per vessel and per patient levels) for functionally significant coronary artery disease with a stress-only protocol compared with the stress/rest protocol
Utility of rest perfusion assessment (2) | 6 weeks
  Sensitivity (per vessel and per patient levels) for functionally significant coronary artery disease with a stress-only protocol compared with the stress/rest protocol
Utility of rest perfusion assessment (3) | 6 weeks
  Specificity (per vessel and per patient levels) for functionally significant coronary artery disease with a stress-only protocol compared with the stress/rest protocol
Subjective experience | 1 week
  Comparison of patient tolerability and experience for each protocol (accelerated CMR, standard CMR and CTCA), as determined by a self-administered questionnaire rating patient comfort, symptoms experienced and perceived scan duration: 4 point scale [1-4 with higher scores meaning worse outcome].
Time duration of each scan/scan component. | 1 week
  Comparison of the time duration of each scan component (accelerated versus standard CMR versus CT protocols).
Image quality | 1 week
  Image quality of each scan/scan component, assessed visually on a 4-point score - excellent (3), good (2), moderate (1) and poor (0).
Cost analysis | 2 years
  A cost consequence and budget impact analysis will be carried out, quantifying the effects of introducing the different diagnostic strategies into the current clinical pathway. Intervention costs and associated healthcare costs will be estimated for each testing strategy. Data on resource use such as staff time, scan duration and hospital days will be collected during the study period. Relevant unit costs will be applied to estimate the total costs. Generalised linear models will be used to analyse the data with adjustments that complement the secondary analyses (above), while accounting for the nature of skewed data. Uncertainty will be estimated by calculating 95% confidence intervals through non-parametric bootstrapping. Scenario-based sensitivity analyses will also be performed and threshold analyses to characterise uncertainty.

CONTACTS AND LOCATIONS:
Overall Officials: Jayanth Arnold, Principal Investigator — University of Leicester
Locations (1):
- Glenfield Hospital, Leicester, Leics, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
no plan at the current time